CLINICAL TRIAL: NCT06127823
Title: Effect of Intensive Nutrition Training, Education, and Support Versus Standard Care in Reducing the Need for Insulin Therapy in Gestational Diabetes (INTENSE-GDM): A Randomised Controlled Trial
Brief Title: Effect of Intensive Nutrition Training, Education, and Support in Gestational Diabetes - The INTENSE-GDM TRIAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Bettina Ewers, Head of Nutrition, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23055674
Record Dates: First submitted 2023-10-30; First posted 2023-11-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: GDM; Gestational Diabetes; Nutritional and Metabolic Diseases; Nutrition Therapy; Medical Nutrition Therapy
Keywords: GDM; Nutrition care; Dietary management; Insulin use; Hospital costs
MeSH Terms: conditions — Diabetes, Gestational; Nutritional and Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: The INTENSE-GDM trial is a randomised controlled parallel group open-label effectiveness trial. Participants will be randomised to either an intensive dietary counselling group or a usual dietary care group (control group) in a 1:1 ratio.
Masking Description: The randomisation list will be made by a researcher/statistician not involved in the trial, who will be the only person to access the randomisation list during the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive dietary care group (Experimental): Women randomised to the intensive dietary intervention group will receive one initial dietary counselling consultation (60 min), and two mandatory follow-up consultations (2 x 30 min) with a dietitian. In addition, participants in this group will be offered 1-2 follow-up consultations (1-2 x 15-30 min) if needed.
  Interventions: Behavioral: Dietary treatment
- Standard dietary care group (Active Comparator): Women randomised to the standard dietary care group will receive one dietary counselling consultation (60 min) according to the initial dietary counselling described without any follow-up consultations with a dietitian. Participants are encouraged to follow their dietary plan until delivery.
  Interventions: Behavioral: Dietary treatment

INTERVENTIONS:
Behavioral: Dietary treatment — Dietary counselling

SUMMARY:
The treatment of gestational diabetes (GDM) primarily revolves around consuming an optimal diet that does not cause blood glucose levels to become excessively high and provides an adequate supply of micro- and macronutrients without resulting in excessive weight gain during pregnancy. In some cases, it may become necessary to supplement with insulin during pregnancy. However, insulin treatment is associated with personal, health-related, and healthcare cost-related implications. The rationale for this study is the lack of knowledge regarding whether the extent of support and guidance from a dietitian during pregnancy has an impact on the treatment outcomes for both the mother and the child in cases of GDM. The overall objective is to investigate differences in clinical, cost-related, and patient-reported outcomes between women with GDM randomised to either intensive dietary therapy or standard dietary care (control). The primary endpoint is the effect of intensive dietary therapy on the likelihood of remaining treated with diet only vs. needing insulin therapy. The study design is a randomised controlled parallel group open-label effectiveness trial including 214 women with GDM.

DETAILED DESCRIPTION:
Gestational diabetes (GDM) is defined as glucose intolerance with onset or first recognition during pregnancy. The disease is characterized by hyperglycaemia and a marked insulin resistance secondary to placental hormonal release. Risk factors for developing GDM in pregnancy include obesity, excessive gestational weight gain, previous GDM, glucosuria, family history of diabetes, ethnicity, and hypertension. Hyperglycaemia is associated with serious short- and long-term complications for mother and child including delivering large-for-gestational-age (LGA) babies, macrosomia, preterm birth, caesarean section, preeclampsia, birth injury, respiratory distress syndrome, neonatal hypoglycaemia, jaundice, and increased admission to neonatal intensive care unit (NICU). First-line treatment in GDM after diagnosis is dietary therapy including a systematic and detailed dietary assessment to identify relevant areas for adjusting the diet and overall lifestyle. The overall goals with dietary therapy are 1) To provide adequate calories and micro- and macronutrients to meet the needs of pregnancy consistent with maintaining normoglycaemia, 1) To improve glycaemic control; and 3) To secure appropriate gestational weight gain and avoid excessive weekly gestational weight gain. Currently, no evidence exists for specific recommendations concerning the optimal frequency, intensity, or duration of visits with a dietitian for improving maternal, foetal, or neonatal outcomes. National clinical guidelines for treatment of GDM recommends up to three visits with a dietitian depending on the time of diagnosis. However, in the latest national clinical guidelines under review this has been changed to only one visit.

In most cases dietary improvements are sufficient to achieve glycaemic goals but around one third of all women with GDM will need insulin therapy at some point during pregnancy. Decision about additional insulin therapy is based on a combination of ultrasound findings and dietary glycemic control as indicated by the blood glucose protocol as assessed by an obstetrician. Insulin therapy can improve glycaemic control and has been shown to be effective in reducing the rate of macrosomia in GDM. But use of insulin during pregnancy is also associated with several clinical implications, increased hospital and medical costs as well as higher costs in relation to delivery, and neonatal care, and personal burden affecting women with GDM.

In summary, the most optimal way to deliver dietary therapy to women with GDM is not known. The possibility that intensive dietary therapy may reduce the need for initiating insulin treatment without increasing hospital service costs for these women in comparison with women receiving standard dietary care needs to be explored.

The overall objective is to investigate the effectiveness and hospital service costs of implementing an intervention with intensive dietary counselling and support during pregnancy in women with GDM.

The INTENSE-GDM trial is a randomised controlled parallel group open-label effectiveness trial including 214 women with GDM. Participants will attend one consultation with a dietitian in the standard care group and up to 5 consultations (including 2 mandatory follow-up visits and 2 optional follow-up visits) with a dietitian in the intensive dietary counselling group. Both groups will receive one end-of-intervention telephone call.

The primary endpoint is the percentage of women with GDM treated with insulin therapy in the intervention group and the control group at delivery. Secondary endpoints include maternal endpoints (changes in body weight from referral to delivery, changes in glycaeted hemoglobin A1c from referral to delivery, time to insulin treatment onset, mean prescribed initial and maximal insulin dose, neonatal endpoints (percentage of LGA, small for gestational age, macrosomia new-borns respectively, percentage of new-borns with neonatal hypoglycaemia and percentage of new-borns admitted to NICU). Descriptive/exploratory endpoints include changes in maternal endpoints (percentage of cases of preeclampsia, preterm births, cases of acute and planned caesarean sections), neonatal endpoints (percentage of cases of neonatal jaundice, questionnaires (diabetes diet-related quality of life, well-being, perceived autonomy support and competence in diet and diabetes, treatment satisfaction and physical activity during pregnancy). Hospital costs will be analysed for the two study groups (intensive dietary therapy vs. standard care) including costs from referral with GDM to discharge after delivery divided into the categories 1) outpatient contacts and costs related to the treatment of GDM, 2) delivery costs, 3) inpatient costs after delivery for mother and offspring separately, including NICU costs and 4) total net costs. Additionally, adherence to intervention (number of no shows for planned visits), number and types of visits (face-to-face, video and telephone), changes in dietary intake and adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed women with GDM referred to Department of Obstetrics Herlev Hospital
* Women diagnosed with GDM based on 2-hour OGTT plasma glucose value ≥ 9.0 mmol/l
* Women diagnosed with GDM based on at least 2 plasma glucose measurements above targets (either pre-prandial ≥6.0 mmol/l, or 2-hours postprandial ≥8.0 mmol/l)
* GA at GDM diagnosis ≤ 34
* Women with an estimated probability of ≥20% for initiating insulin treatment during pregnancy. The estimated probability is based on a logistic regression model developed at SDCC and includes the following variables: prepregnancy BMI, GA at GDM diagnosis, and HbA1c at GDM diagnosis. In cases where HbA1c has not been measured during the initial visit with the dietitian (screening visit), prepregnancy BMI, GA at the time of diagnosis and 2H OGTT will be used to estimate the probability of initiating insulin therapy.
* Provided voluntary written informed parental consent in Danish or English or after translation by an interpreter for non-Danish and non-English speaking parents

Exclusion Criteria:

* Bariatric surgery
* Other intercurrent illness (e.g., cancer, ulcerative colitis) as judged by medical experts
* Uncontrolled medical issues, as judged by medical experts
* Concomitant participation in other clinical trials that could interfere with the INTENSE- GDM Trial as evaluated by the principle investigator
* Unable to understand the informed consent/procedures regardless of spoked language

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only biological gender
Enrollment: 214 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of insulin-treated | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Percentage of women with GDM treated with insulin therapy in the two study groups

SECONDARY OUTCOMES:
Maternal body weight | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Changes in body weight, kg
Maternal glycaemic control | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Changes in maternal HbA1c, mmol/mol
Onset of insulin treatment | From date of randomisation until date of first insulin prescription, assessed from study completion up to 24 weeks
  Time to insulin treatment onset, days
Prescribed insulin | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Mean prescribed initial and maximal insulin dose, units/kg body weight
Large for gestational age (LGA) | At delivery, assessed from study completion up to 24 weeks
  LGA new-borns, %
Small for gestational age (SGA) | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  SGA new-borns, %
Macrosomia (birth weight >4,500 g) | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Newborns with macrosomia, %
Neonatal hypoglycaemia | From date of randomisation until data of discharge after child delivery, assessed from study completion up to 24 weeks
  New-borns with neonatal hypoglycaemia, %
Admission to neonatal intensive care unit (NICU) | From date of randomisation until data of discharge after child delivery, assessed from study completion up to 24 weeks
  New-borns admitted to NICU, %

OTHER OUTCOMES:
Neonatal jaundice | From date of randomisation until data of discharge after child delivery, assessed from study completion up to 24 weeks
  Newborns with neonatal jaundice, n (%)
Planned caesarean sections | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Cases of planned caesarean sections, n (%)
Acute caesarean sections | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Cases of acute caesarean sections, n (%)
Preterm births | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Cases of preterm births, n (%)
Preeclampsia | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Cases of preeclampsia, n (%)
Diabetes Diet-related Quality of Life (DDQOL) | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Changes in DDQOL, total score
Well-being (WHO-5) | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Changes in WHO-5, total score
Health Care Climate Questionnaire (HCCQ) | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Changes in HCCQ, total score
Perceived Competence in Diabetes Scale (PCDS) | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Changes in PCDS, total score
Pregnancy Physical Activity Questionnaire (PPAQ) | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Changes in PPQA, total score
Treatment satisfaction | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Treatment satisfaction, categorical distribution of answers
Adherence to intervention | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  No shows for planned visits, n (%)
Type of visits to the dietitian | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Face-to-face, video and telephone, n (%)
Changes in dietary intake with focus on carbohydrate intakes (total intake and meals) | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Based on an interview
Adverse events | From date of randomisation until date of child delivery, assessed from study completion up to 24 weeks
  Type of adverse events described
Outpatient contacts | From date of randomisation until date of discharge after child delivery, assessed from study completion up to 24 weeks
  Number and type of contacts at hospital related to pregnancy and diabetes treatment, n (%)
Outpatient costs related to the treatment of GDM from referal until | From date of randomisation until date of discharge after child delivery, assessed from study completion up to 24 weeks
  Diagnosis-related rates, DKK
Delivery costs | From date of labour until date of child delivery, assessed from study completion up to 24 weeks
  Diagnosis-related delivery costs, DKK
Inpatient costs after delivery for the mother | From data of child delivery until date of discharge after child delivery, assessed from study completion up to 24 weeks
  Impatient costs after delivery related to admission to a neonatal intensive care unit, DKK
Inpatient costs after delivery for the offspring | From data of child delivery until date of discharge after child delivery, assessed from study completion up to 24 weeks
  Inpatient costs after delivery related to admission to a neonatal intensive care unit, DKK
Total net costs | From date of randomisation until date of discharge after child delivery, assessed from study completion up to 24 weeks
  Total costs including GDM- and pregnancy-related hospital cost and medical costs, DKK

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Ewers, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ewers B, Blond MB, Kelstrup L, Foghsgaard S, Bergholt T, Hansen MJ, Storgaard H, Holmager P, Mathiesen ER. Effect of intensive nutrition training, education and support versus standard therapy in reducing the need for insulin therapy in gestational diabetes (INTENSE-GDM): a protocol for a randomised controlled single-centre trial in Denmark. BMJ Open. 2025 Feb 17;15(2):e089231. doi: 10.1136/bmjopen-2024-089231. PMID 39961720

DOCUMENTS (1):
  • Study Protocol (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT06127823/Prot_002.pdf